CLINICAL TRIAL: NCT07223918
Title: Pilot Testing for a Personalized Decision-Aid to Guide Tracheostomy and Prolonged Mechanical Ventilation Decision-Making
Brief Title: Personalized Decision-Aid to Guide Tracheostomy and Prolonged Mechanical Ventilation Decision-Making
Status: Completed | Type: Observational
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 23-0171; K23HL141704 (NIH)
Record Dates: First submitted 2025-10-29; First posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Acute Respiratory Failure; Mechanical Ventilation; Tracheostomy
Keywords: acute respiratory failure; prolonged mechanical ventilation; tracheostomy; shared decision-making

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surrogates: Surrogate decision-makers are individuals who the primary medical team has determined to be the decision-maker for incapacitated patients on ventilators. Surrogates will be asked to review TRACH-Support if the patient has been receiving mechanical ventilation for >7 days or has been asked to consider a tracheostomy.
  Interventions: Behavioral: TRACH-Support
- Healthcare Team Members: Healthcare team members will include critical care and palliative care physicians, APPs, nurses, and respiratory therapists who work in critical care units and routinely engage in discussions with surrogates about tracheostomy and prolonged mechanical ventilation.
  Interventions: Behavioral: TRACH-Support

INTERVENTIONS:
Behavioral: TRACH-Support — TRACH-Support is a newly developed personalized online decision-support tool designed to support shared decision-making for tracheostomy and prolonged mechanical ventilation decision-making (https://www.patientdecisionaid.org/trachsupport/introduction/).

SUMMARY:
The goal of this study is to determine the Usability and Acceptability of a personalized online decision support tool for patients, families, and providers considering long-term breathing support options for patients who cannot breathe by themselves. The tool is called TRACH-Support. The key questions are:

1. Is TRACH-Support usable and acceptable to people who make decisions for patients on breathing machines.
2. Is TRACH-Support usable, acceptable, appropriate, and feasible for medical providers, nurses, and respiratory therapists who care for patients on breathing machines.

In this study, family members of patients on a breathing machine and members of the medical team will review the tool and fill out an online survey describing their thoughts about the tool. A subgroup of individuals who fill out the survey will also be asked to participate in qualitative interviews about their experience with the tool.

DETAILED DESCRIPTION:
This study is primarily designed to assess the Usability and Acceptability of TRACH-Support, a personalized online decision support tool for tracheostomy and prolonged mechanical ventilation, among surrogate decision makers, physicians, advanced practice providers (APPs), nurses, and respiratory therapists. The secondary aim of this study is to determine Appropriateness and Feasibility of implementing TRACH-Support in critical care settings among the healthcare team (physicians, APPs, nurses, and respiratory therapists) and to determine preliminary efficacy at reducing Decisional Conflict among surrogates who use TRACH-Support as compared to historical controls.

The investigators will present TRACH-Support to the above mentioned groups and have them fill out online surveys describing their experience and thoughts with TRACH-Support. A subgroup of individuals will be asked to participate in qualitative interviews to dive deeper into the experience with TRACH-Support and explore potential adaptations prior to wider scale testing.

ELIGIBILITY:
Inclusion Criteria:

Surrogates

* Age >18 years
* English or Spanish speaking
* Surrogate decision-maker for a patient who has been receiving mechanical ventilation for greater than or equal to 7 days or in whom a tracheostomy discussion is planned. The role of surrogate decision-maker will be determined by the medical team (can be either a medical decision power of attorney (MDPOA) or proxy decision-maker).
* As many decisions are made by a group of surrogates rather than a single surrogate, up to 3 surrogates per patient will be enrolled.

Healthcare Team Members

* Age > 18 years
* A critical care or palliative care physician (MD/DO), advanced practice provider (APP), nurse, or respiratory therapist who routinely engages in tracheostomy and PMV discussions

Exclusion Criteria:

Surrogates

* Age < 18 years
* Non-English or Non-Spanish speaking
* Prisoner

Healthcare Team Members

* Age < 18 years
* refuses to evaluate TRACH-Support
* refuses to discuss alternatives to tracheostomy with families

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will focus on 2 broad groups. Surrogates - Almost all patients receiving mechanical ventilation lack decisional capacity. Therefore, all key medical decisions are made by surrogate decision-makers including decisions related to tracheostomy and PMV. We will recruit surrogate decision-makers identified by the primary medical team to evaluate TRACH-Support for patients who have received MV for 7 days or more or for whom a tracheostomy discussion is planned.
  Healthcare Team Members - early qualitative data indicates that decision-making often involves the entire healthcare team. Therefore, we will recruit providers, nurses, and respiratory therapists routinely involved in the care of patients receiving MV to evaluate TRACH-Support.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
System Usability Scale | Baseline
  The System Usability Scale is a 10-item questionnaire using a 5-level Likert scale designed to assess the usability of systems and interventions. The score ranges from 0-100 with higher numbers indicating greater usability.

SECONDARY OUTCOMES:
Acceptability of Intervention Measure | Baseline
  The Acceptability of Intervention Measure (AIM) is a 4 item measure scored on a 5 point Likert scale designed to assess the acceptability of an intervention to a target population. The cumulative score ranges from 4-20. The mean score for all 4 questions for each individual (ranging from 1-5) is also used frequently. In both situations, higher numbers indicate greater Acceptability.
Feasibility of Intervention Measure | Baseline
  The Feasibility of Intervention Measure (FIM) is 4 item measure scored on a 5 point Likert scale designed to assess the feasibility of implementing a new intervention to a target population. The cumulative score ranges from 4-20. The mean score for all 4 questions for each individual (ranging from 1-5) is also used frequently. In both situations, higher numbers indicate greater Feasibility. This outcome was only assessed among members of the healthcare team.
Intervention Appropriateness Measure | Baseline
  The Intervention Appropriateness Measure (IAM) is a 4 item measure scored on a 5 point Likert scale designed to assess the whether an intervention is appropriate in a given context. The cumulative score ranges from 4-20. The mean score for all 4 questions for each individual (ranging from 1-5) is also used frequently. In both situations, higher numbers indicate greater Appropriateness. This measure was only assessed among members of the healthcare team.
Decisional Conflict Scale (low literacy) | Baseline
  The Decisional Conflict Scale (DCS) is a 10-item questionnaire that assess the conflict an individual experiences with a given decision. Each question offers the responses Yes, No, and Unsure. The DCS score ranges from 0-100 with higher numbers indicating greater decisional conflict. The low literacy scale has been validated for individuals with limited reading or response skills. The DCS is the most common outcome assessed in shared decision-making trials. DCS was only assessed among surrogates.

CONTACTS AND LOCATIONS:
Locations (1):
- Denver Health and Hospital Authority, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
As an observational study we do not plan on sharing individual participant data outside of the research team other than de-identified quotes from qualitative interviews.

REFERENCES:
- See also: TRACH-SUpport — https://www.patientdecisionaid.org/trachsupport/introduction/